CLINICAL TRIAL: NCT00988988
Title: The Effects of Ethyl-alpha-Guanido-methyl Ethanoate on Skin Reactions Form Glatiramer Acetate
Brief Title: The Effects of Ethyl-Alpha-Guanido-Methyl Ethanoate on Skin Reactions From Glatiramer Acetate Injections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not approved by IRB
Sponsor: University of Nebraska (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0399-09-FB
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; AGEE; histamine response
MeSH Terms: conditions — Multiple Sclerosis | interventions — Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Steroid Cream (Active Comparator): 1% steroid cream
  Interventions: Drug: 1% Steroid Cream
- AGEE cream (Active Comparator): AGEE cream is a creatine ethyl ester based product (an amino acid) that can be purchased over-the-counter without a prescription and is not FDA controlled
  Interventions: Drug: AGEE cream
- placebo (Active Comparator): inactive cream
  Interventions: Drug: topical placebo cream with no active ingredients

INTERVENTIONS:
Drug: AGEE cream — AGEE cream is a creatine ethyl ester based product (an amino acid) that can be purchased over-the-counter without a prescription and is not FDA controlled. It will be used immediately after injection and repeated as needed.
  Other Names: creatine ethyl ester based topical
  Arms: AGEE cream
Drug: 1% Steroid Cream — comparing to AGEE cream or placebo. 1% steroid cream is available over the counter. To be used immediately after injection and as needed.
  Other Names: generic
  Arms: Steroid Cream
Drug: topical placebo cream with no active ingredients — Cream to be applied immediately after injection and repeated as needed.
  Other Names: generic
  Arms: placebo

SUMMARY:
Participants with multiple sclerosis that are currently treated with glatiramer acetate (GA, Copaxone®) injections and have redness, pain, swelling, itching or a lump at the injection site will be recruited to examine histamine response of three topical treatments to reduce these symptoms.

DETAILED DESCRIPTION:
Participants are asked to be in this study because they have multiple sclerosis, are currently treated with glatiramer acetate (GA, Copaxone®) injections and have redness, pain, swelling, itching or a lump at the injection site.

The purpose of this study is to determine if the use of ethyl-a-guanida-methyl ethanoate (AGEE) will decrease histamine response measured by redness, swelling, and itch response following subcutaneous injection of glatiramer acetate (GA) for the treatment of Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Between ages 19-65
* Laboratory supported diagnosis of multiple sclerosis
* Currently treated with injectable GA, experiencing wheal and flare after injection

Exclusion Criteria:

* Unable to give informed consent
* Treated with any other therapy for Multiple Sclerosis

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02 (Estimated); Primary Completion 2012-08-03 (Actual); Study Completion 2012-08-03 (Actual)

PRIMARY OUTCOMES:
Histamine response after ethyl-α-guanida-methyl ethanoate (AGEE) and subcutaneous injection of glatiramer acetate | Three weeks
  To determine if the use of ethyl-α-guanida-methyl ethanoate (AGEE) will decrease histamine response measured by wheal, flare and itch response following subcutaneous injection of glatiramer acetate for the treatment of Multiple Sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Mary Filipi, PhD, APRN, Principal Investigator — University of Nebraska